CLINICAL TRIAL: NCT02881073
Title: PARROT Ireland: Placental Growth Factor in Assessment of Women With Suspected Pre-eclampsia to Reduce Maternal Morbidity: a Randomised Control Trial
Brief Title: Placental Growth Factor Assessment of Women With Suspected Pre-eclampsia
Acronym: PARROT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Irish Centre for Fetal and Neonatal Translational Research (Other)
Collaborators: National Maternity Hospital, Ireland (Other); Rotunda Maternity Hospital, Dublin (Unknown); Coombe Women and Infants University Hospital (Other); University College Hospital Galway (Other); Royal Jubilee Maternity Hospital, Belfast (Unknown); Cork University Maternity Hospital (Other); Univerisy Maternity Hospital, Limerick (Unknown); University College Cork (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Diagnostic
Other Study IDs: LK001-16
Record Dates: First submitted 2016-08-10; First posted 2016-08-26 (Estimated); Last update posted 2019-08-07 (Actual); Status verified 2019-08

CONDITIONS: Pre-eclampsia; Pregnancy, High Risk; Pregnancy Complications
Keywords: Placental Growth Factor; Maternal Morbidity; Neonatal Morbidity; Pre-eclampsia; Heath Economics
MeSH Terms: conditions — Pre-Eclampsia; Pregnancy Complications

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): Eligible women at participating centres prior to roll-out of PlGF testing (as per stepped wedge trial design) will be managed according to HSE/Institute of Obstetrician and Gynaecologists' National Guidelines for 'The management of hypertensive disorders during pregnancy' & "The management of Pre-eclampsia" or by NICE guidelines for "Management of Hypertension in Pregnancy" for those in Northern Ireland.
- Maternal plasma PlGF quantification (Active Comparator): Women in the interventional arm will have an additional point of care test performed at the time of enrolment for immediate PlGF quantification. The PlGF measurement will be reported as the absolute value in pg/ml with the following ranges given:
  * PlGF <12 pg/ml: Very low
  * PlGF ≥12 and <100 pg/ml: Low
  * PlGF ≥100 pg/ml: Normal
  All hospitals will follow National Guidelines for 'The management of hypertensive disorders during pregnancy' & "The management of Pre-eclampsia" with the additional integration of PlGF results as indicated in the algorithm.
  Interventions: Other: Maternal plasma PlGF quantification

INTERVENTIONS:
Other: Maternal plasma PlGF quantification — A point of care test performed on maternal plasma, to quantify the level of the protein PlGF (placental growth factor) in the serum of the pregnant woman with suspected pre eclampsia to help the clinician in stratifying the level of further care for her in her pregnancy
  Arms: Maternal plasma PlGF quantification

SUMMARY:
The primary aim is to establish the effectiveness of plasma PlGF measurement in reducing maternal morbidity (with assessment of perinatal safety in parallel) in women presenting with suspected pre-eclampsia prior to 37 weeks' gestation.

The long term aim is to demonstrate that knowledge of PlGF measurement enables appropriate stratification of the antenatal management of women presenting with suspected pre-eclampsia, such that those at highest risk receive greater surveillance with a decrease in maternal adverse outcomes, and those at lower risk can be managed without unnecessary admission and other interventions, such that the results would influence international clinical practice in antenatal patient healthcare

DETAILED DESCRIPTION:
Pre-eclampsia (PET), a disease of late pregnancy characterised by hypertension and proteinuria, complicates 2-8% of pregnancies and is associated with significant maternal and neonatal morbidity and mortality. Many reports have highlighted the frequent substandard care, often attributed to clinicians not identifying the seriousness of clinical signs suggestive of the disease. Consequently, improvements in prediction of development of PET have the potential to vastly improve clinical outcomes and reduce costs.

Placental Growth Factor (PlGF) belongs to the vascular endothelial growth factor (VEGF) family and represents a key regulator of angiogenic events in pathological conditions. PlGF exerts its biological function through the binding and activation of the receptor Flt-1. In PET, it is thought that endothelial dysfunction leads to an increased level of a circulating decoy receptor, known as soluble Flt-1, (sFlt-1), a soluble receptor for both VEGF-A and PlGF.

In 2013, the INFANT team were part of an international group that published the first multicentre prospective study (PELICAN) evaluating the use of PlGF in women presenting with suspected PET, which reported high sensitivity (95-96%) and negative predictive value (95-98%) for low PlGF in determining need for delivery for confirmed PET within 14 days. This study suggests that PlGF testing presents a realistic and innovative adjunct to the management of women with suspected PET, especially those presenting preterm.

ELIGIBILITY:
Inclusion Criteria:

Pregnant women between 20+0 and 36+6 weeks of gestation (inclusive) Singleton pregnancy Aged 18 years or over Able to give informed consent, presenting with any symptoms of suspected pre-eclampsia

* Headache
* visual disturbances
* epigastric or right upper quadrant pain
* increasing oedema
* hypertension
* dipstick proteinuria
* suspected fetal growth restriction
* if the healthcare provider deems that the woman requires evaluation for possible pre-eclampsia

Exclusion Criteria:

* Confirmed pre-eclampsia at point of enrolment (sustained hypertension with systolic BP ≥ 140 or diastolic BP ≥ 90 on at least two occasions at least 4hrs apart) with significant quantified proteinuria (>300mg protein on 24hr collection, urine protein creatinine ratio >30mg/mmol or +3 Dipstick Proteinuria)
* >37 weeks gestation
* Abnormal PET bloods
* Multiple pregnancy at any time point
* Decision regarding delivery already made
* Lethal fetal abnormality
* Previous participation in PELICAN trial in a prior pregnancy
* Unable/unwilling to give informed consent

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2313 (Actual)
Dates: Start 2017-06-29 (Actual); Primary Completion 2019-04-26 (Actual); Study Completion 2019-04-26 (Actual)

PRIMARY OUTCOMES:
Maternal Morbidity | up to 6 weeks post delivery
  assessed using a composite outcome combining the modified fullPIERS model for pre-eclampsia with sustained systolic blood pressure ≥ 160 mmHg
Neonatal Morbidity | From neonates birth until time of discharge from the neonatal unit/hospital, up to 6 weeks post delivery
  assessed using a composite neonatal score

SECONDARY OUTCOMES:
Maternal Morbidity | up to 6 weeks post delivery
  Final diagnosis of hypertensive disorder of pregnancy
Maternal Morbidity | up to 6 weeks post delivery
  Maternal morbidity by fullPIERS model (without systolic hypertension)
Maternal Outcome- | up to 6 weeks post delivery
  Progression to severe pre-eclampsia as defined by ACOG
Maternal Outcome | up to 6 weeks post delivery
  Caesarean section: emergency or elective
Maternal Outcome | up to 6 weeks post delivery
  Elective delivery: induction of labour or Caesarean section
Fetal Outcome | up to 6 weeks post delivery
  Gestation at diagnosis of pre-eclampsia
Fetal Outcome | up to 6 weeks post delivery
  Fetal growth restriction identified on antenatal ultrasound
Fetal Outcome | up to 6 weeks post delivery
  Gestation at delivery
Heath Economic Outcomes | up to 6 weeks post delivery
  Costs to Health Service of Community Based care: assessed through chart review at discharge
Heath Economic Outcomes | up to 6 weeks post delivery
  Costs to Health Service of inpatient/day case care: Assessed by chart review at discharge thought HIPE/HPO/Length of stay for both mother and baby
Fetal Quality of Life Assessment | up to 6 weeks post delivery
  Use utility values / decrements scale for infants to estimate the cost effectiveness of the intervention
Heath Economic Outcomes -Transport costs to patient of appointments | up to 6 weeks post delivery
  Identified through a costing questionnaire given to the patient to complete at discharge from hospital post delivery. Will ask how far patient lives from their GP and their hospital and their means of transport when attending appointments and thus calculate the transport cost to a patient throughout the pregnancy of attending their appointments.
Maternal Quality of Life | Assessed at two individual timepoints during the trial: once at time of enrolment to the study and repeated again post delivery and up to 6 weeks post delivery
  Assessed through EQ-5D-5L questionnaire
Maternal Quality of Life | Assessed at two individual timepoints during the trial: once at time of enrolment to the study and repeated again post delivery and up to 6 weeks post delivery
  Assessed through SF-6D questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Louise C Kenny, PhD, MD, Principal Investigator — Irish Centre for Fetal and Neonatal Translational Research
Locations (7):
- Ireland (7):
  - Royal Jubilee Maternity Hospital, Belfast
  - Cork University Maternity Hospital, Cork
  - Coombe Womens & Infants University Hospital, Dublin
  - National Maternity Hospital, Dublin
  - Rotunda Maternity Hospital, Dublin
  - University College Hospital Galway, Galway
  - University Maternity Hospital Limerick, Limerick

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hayes-Ryan D, Khashan AS, Hemming K, Easter C, Devane D, Murphy DJ, Hunter A, Cotter A, McAuliffe FM, Morrison JJ, Breathnach FM, Dempsey E, Kenny LC, O'Donoghue K; PARROT Ireland trial group. Placental growth factor in assessment of women with suspected pre-eclampsia to reduce maternal morbidity: a stepped wedge cluster randomised control trial (PARROT Ireland). BMJ. 2021 Aug 13;374:n1857. doi: 10.1136/bmj.n1857. PMID 34389547
- [Derived] Hayes-Ryan D, Meaney S, Nolan C, O'Donoghue K. An exploration of women's experience of taking part in a randomized controlled trial of a diagnostic test during pregnancy: A qualitative study. Health Expect. 2020 Feb;23(1):75-83. doi: 10.1111/hex.12969. Epub 2019 Oct 2. PMID 31578808
- [Derived] Hayes-Ryan D, Hemming K, Breathnach F, Cotter A, Devane D, Hunter A, McAuliffe FM, Morrison JJ, Murphy DJ, Khashan A, McElroy B, Murphy A, Dempsey E, O'Donoghue K, Kenny LC. PARROT Ireland: Placental growth factor in Assessment of women with suspected pre-eclampsia to reduce maternal morbidity: a Stepped Wedge Cluster Randomised Control Trial Research Study Protocol. BMJ Open. 2019 Mar 1;9(2):e023562. doi: 10.1136/bmjopen-2018-023562. PMID 30826791